CLINICAL TRIAL: NCT06125938
Title: Comparative Study Between Autogenous Bone Block and Tent Pole Technique for Augmentation of Atrophic Anterior Maxilla A Randomized Clinical Trial
Brief Title: Comparative Study Between Autogenous Bone Block and Tent Pole Technique for Augmentation of Atrophic Anterior Maxilla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Youmna Mohamed Mahmoud Hassan Abdelhady, master candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 40723
Record Dates: First submitted 2023-10-27; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Bone Atrophy, Alveolar
Keywords: bone augmentation ,tent pole
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tent pole technique (Experimental): The screw tent-pole method is an effective technique to achieve initial reconstruction of alveolar bone deficiencies
  Interventions: Procedure: tent pole technique
- autogenous bone block technique (Active Comparator): Bone block graft has been the gold standard for restoring deficient regions.
  Interventions: Procedure: Autogenous bone block technique

INTERVENTIONS:
Procedure: tent pole technique — The screw tent-pole method is an effective technique to achieve initial reconstruction of alveolar bone deficiencies
  Arms: tent pole technique
Procedure: Autogenous bone block technique — Bone block graft has been the gold standard for restoring deficient regions.
  Arms: autogenous bone block technique

SUMMARY:
The goal of this clinical trial is to compare in patients with atrophied anterior maxilla, bone augmentation techniques ( gold standard bone block and tent pole technique).

The main question it aims to answer is :

Does screw tent pole technique provides better bone gain than autogenous bone block in atrophied anterior maxilla?

* primary objective to assess amount of bone gain
* secondary objective assess bone quality Participants will be randomly divided into two groups study group ( tent pole technique) and control group ( bone block) - each group will be followed up monthly for soft tissue dehiscence and after 6 month to assess bone gain and bone quality and then implant placement.

DETAILED DESCRIPTION:
• Research question: Does screw tent pole technique provides better bone gain than autogenous bone block in atrophied anterior maxilla?

• Rationale for conducting the research: Several methods have been developed for the augmentation of the deficient bone volume. These include Guided Bone Regeneration (GBR) with barrier membranes, onlay bone grafting, ridge splitting and distraction osteogenesis.

The screw tent-pole method is an effective technique to achieve initial reconstruction of alveolar bone deficiencies. Previous studies have proven that screw tent pole technique is recommended in reconstruction of atrophied alveolar bone and its good outcome in contrary to other bone graft techniques.

This study aim to compare the outcome of screw tent pole technique to conventional gold standard technique of block bone grafts in atrophied anterior maxilla.

• Primary and secondary objectives:

* primary objective to assess amount of bone gain
* secondary objective assess bone quality . Trial design: Randomized clinical trial, Unicentered, Parallel groups, 2 arms, Allocation ratio 1:1, Equivalent trial • PICO: Population: patients with atrophied Anterior Maxillary area (with initial ridge width of ≤ 5 mm and moderate bone height) Intervention: Screw Tent-Pole technique Control group: Autogenous Bone Block technique Outcome: bone gain , histomorphometric evaluations, dehiscence.

  * Interventions

    * Surgical Protocol

A. Screw Tent pole technique

* A prophylactic antibiotics administration was conducted.
* All surgical procedures were performed under local anesthesia.
* A trapezoid incision will be formed to expose the edentulous alveolar ridge in recipient site.
* A full-thickness flap will be retracted to expose the alveolar bone. 5
* Titanium screws (1.5 mm) will be placed perpendicular to alveolar bone so that approximately 5 to 7 mm of screw threat will be exposed.
* A posterior releasing incision was made over ramus to provide access to the donor site.
* Autogenous bone graft taken from donor site area using ACM bur
* The autogenous particles obtained from the donor site will be mixed with xenograft in a 50/50 ratio.
* PRF membrane is then prepared ( PRF membrane formed by withdrawing blood sample from patient into a tube , the tube will be transferred to centrifuge machine -2500 RPM for 10 minutes) and is pierced through the healing abutment and used to cover the bone graft to accelerate wound healing by preventing soft tissue ingrowth.
* A tension-free suture will be completed.
* After 6 months of healing:

A full-thickness flap is retracted to expose the alveolar bone (augmented site).

The screw will be removed, Histopathological biopsy sample of bone will be taken using trephine bur (the same size as pilot drill) and sequential drilling will be done for implant placement at the same visit.

B. Autogenous bone block technique

* A prophylactic antibiotics administration was conducted.
* All surgical procedures were performed under local anesthesia.
* A trapezoid incision will be formed to expose the edentulous alveolar ridge in recipient site.
* A full-thickness flap will be retracted to expose the alveolar bone.
* A posterior releasing incision was made over ramus to provide access to the donor site.
* The size of the ramus graft will be determined from the recipient site, and bone osteotomy of cortical and cancellous bone will be done by Piezo-electric bone surgery.
* The outlined graft was mobilized from its bed using chisels and the bone block will be placed in defected anterior maxilla and stabilized using micro screws.
* particulate Autogenous bone graft will also be taken from donor site area using ACM bur and mixed with xenograft in a 50/50 ratio and then placed to fill the space in between the bone block.
* PRF membrane is then prepared ( PRF membrane formed by withdrawing blood sample from patient into a tube , the tube will be transferred to centrifuge machine -2500 RPM for 10 minutes) and is pierced through the healing abutment and used to cover the bone graft to accelerate wound healing by preventing soft tissue ingrowth.
* A tension-free suture will be completed.
* After 6 months of healing:

A full-thickness flap is retracted to expose the alveolar bone (augmented site).

The screw will be removed, Histopathological biopsy sample of bone will be taken using trephine bur (the same size as pilot drill) and sequential drilling will be done for implant placement at the same visit.

• Post-operative care:

* Avoid traumatization of the surgical site.
* Patients must abstain from brushing the surgical area. Instead, a disinfecting mouth rinse should be used (e.g. chlorhexidine 0.2%).
* ·Instruct the patient not to touch or manipulate the surgical area.
* ·Ice packs for 10 minutes every 30 minutes for 24 hours.
* Do not use removable dentures during the expansion phase. Temporary fixed partial dentures must be adjusted to the expected tissue gain.
* ·No consume of tobacco
* ·Post-operative medications will be prescribed as follows:
* Amoxicillin/clavulanic acid tablets 10mg/kg every 12 hours for 7 days, diclofenac potassium 50mg every 8 hours for 4 days and then as needed, metronidazole 5 mg/kg every 8 hours for 7 days and chlorhexidine gluconate
* 0.1% mouthwash 3 times daily for 14 days.

Clinical follow up:

-The dehiscence will be followed up every month.

Radiographic follow up:

-Immediately after surgery and after six months, CBCT will be obtained to evaluate bone gain in each group

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy patients (American Society of Anesthesiologists -ASA I and II); older than 18 years
* Patients with atrophic anterior maxilla ,with initial ridge wi¬dth of ≤ 5 mm and moderate bone height as diagnosed at the time of digital implant planning
* No intraoral soft and hard tissue pathology.
* Cone Beam Computer Tomography scan before and after bone augmentation.
* Apprehensive to be in the study

Exclusion Criteria:

* Bad oral hygiene.
* smokers (>10 cigarettes/day);
* Existence of a bone metabolic disease; currently taking drugs that might influence bone metabolism
* Radiotherapy or chemotherapy for malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Bone Gain | 6 month
  to assess amount of bone gain before and after 6 month of the surgical procedure

SECONDARY OUTCOMES:
Bone quality evaluation | 6 month post-operative
  the bone quality through bone core biopsy by trephine bur will be evaluated in the two techniques after 6 months post-operative

OTHER OUTCOMES:
soft tissue dehiscence | monthly for 6 months post-operative
  the soft tissue around the surgical site will be evaluated periodically through clinical inspection for 6 months post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Youmna M Abdelhady, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt